CLINICAL TRIAL: NCT02167828
Title: Increasing Social Support to Improve HIV Care Engagement and Adherence
Brief Title: Increasing Social Support to Improve HIV Care Engagement and Adherence in St. Petersburg, Russia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00021451; R21MH102193 (NIH)
Record Dates: First submitted 2014-05-01; First posted 2014-06-19 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: HIV; AIDS
Keywords: HIV; AIDS; treatment adherence; social network
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Support (Experimental): Participants will be trained to give one another ongoing, theory-based but personally-tailored advice, recommendations, and support to encourage entry to HIV medical care, remaining in care, and adhering to medication regimens when they are prescribed. The intervention's intent is to increase mutual support, positive attitudes, intentions, plans, and collective self-efficacy for care engagement.
  Interventions: Behavioral: Social Support
- No Intervention (No Intervention): Participants in this arm will not receive an intervention.

INTERVENTIONS:
Behavioral: Social Support
  Other Names: Social Network Training
  Arms: Social Support

SUMMARY:
Prior research has documented serious health, mental health, and social-behavioral issues among people living with HIV (PLH) in St. Petersburg. The investigators have established that PLH are clustered in friendship groups with other HIV+ persons and that an intervention delivered to groups composed of HIV+ men who have sex with men (MSM) who were friends in real life reduced mental health distress more than individual counseling. Specific aims of the collaborative mixed-methods, qualitative/ quantitative research are to: (1) identify facilitators and barriers of medical care attendance and ART adherence among PLH in St. Petersburg; (2) integrate these data into an intervention designed to increase HIV care attendance, retention, and adherence; (3) carry out a test-of-concept pilot study that recruits groups of PLH friends and delivers an intervention to intact PLH friendship groups to encourage mutual social support for attending medical appointments and adhering to HIV care; and (4) evaluate the effects of the intervention on both behavioral and biological measures, including viral load. These specific aims will be achieved by research carried out in two phases:

In Phase I, we will conduct in-depth interviews with 60 PLH and key informants in St. Petersburg purposively selected to include HIV+ persons in and not in medical care, adherent or not adherent to ART, and including men and women representing diverse exposure risks. In-depth interviews will be analyzed to identify factors associated with attending or not attending care and adhering or not adhering to ART, as well as identifying how HIV+ friends can support one another in HIV care entry, retention, and adherence.

In Phase II, the investigators will undertake a randomized intervention pilot study in which 20 groups of PLH friends are recruited by enrolling a PLH seed who is not reliably in care or is ART nonadherent and then recruiting all friends known by the seed to also be HIV+. A 7-session group intervention will be undertaken with all members of the friendship groups in the experimental condition to increase care and adherence-related social support, problem-solving, and mutual assistance for care. Baseline to 6-month followup data will determine whether the intervention produces greater improvement than found in the comparison group in care attendance and treatment adherence, improved mental health, lower substance use, and lower HIV viral load.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Self-report as being HIV-positive
* Except for initial seeds, must be named by an already-enrolled participant as an HIV-positive friend
* Do not plan to move from the St. Petersburg area for the next 12 months
* Able to provide written informed consent and do not exhibit severe alcohol intoxication, drug use impairment, or acute psychiatric impairment.

Exclusion Criteria:

* Age 17 or younger
* Self-report as HIV-negative
* Not named as an HIV-positive friend by an already-enrolled participant
* Plans to move from the St. Petersburg area in the next 12 months
* Exhibit severe alcohol intoxication, drug use impairment, or acute psychiatric impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Number of Medical Appointments Attended | 6 months
  measure--through self-report--the number of medical appointments each participant attends in a six-month period.

SECONDARY OUTCOMES:
Number of Prescribed Antiretroviral Medication Doses Taken | 6 months
  measure--through self-report--the number of medication doses each participant takes in a six-month sample.
CD4 Level | 6 months
  Viral load (i.e., CD4 level) in each participant will be measured via blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Kelly, PhD, Principal Investigator — Medical College of Wisconsin; Yuri A. Amirkhanian, PhD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- Center for AIDS Intervention Research, Medical College of Wisconsin, Milwaukee, Wisconsin, United States
- Botkin Hospital for Infectious Diseases #30, Saint Petersburg, Russia